CLINICAL TRIAL: NCT00889655
Title: A Prospective, Randomized Controlled Trial Comparing the Efficacy and Patient Tolerability of MiraLAX (PEG 3350) vs Golytely as Bowel Preparation for Screening Colonoscopy
Brief Title: A Trial Comparing Bowel Preparation and Patient Tolerability of Miralax Versus Golytely
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Glenn Eisen, Oregon Health & Science University, Division of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00005072
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Colonoscopy
Keywords: efficacy of bowel cleansing; patient tolerability; Golytely; MiraLax; colonoscopy preparation; bowel preparation; screening colonoscopy
MeSH Terms: interventions — Golytely; Polyethylene Glycols; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Golytely (Active Comparator): 216 patients at random will provided a prescription for the standard 4 L golytely preparation as the bowel cleanser for their colonoscopy
  Interventions: Drug: Golytely (polyethylene glycol)
- MiraLax (Experimental): 216 patients will be randomized to take 238 gm of miralax mixed with 64 oz of gatorade for their bowel cleanser
  Interventions: Drug: MiraLax (polyethylene glycol 3350)

INTERVENTIONS:
Drug: Golytely (polyethylene glycol) — 4 L of golytely, in split dosing. If the patient has a morning colonoscopy, they will take 2 L of golytely over 2 hours the morning prior to their procedure and repeat this at 6 pm the night prior to their procedure.
  Arms: Golytely
Drug: MiraLax (polyethylene glycol 3350) — 238 gm of MiraLax mixed in 64 oz of Gatorade, to be consumed in split dosing the day prior to scheduled colonoscopy.
  Arms: MiraLax

SUMMARY:
Prior to colonoscopies, the colon is cleansed using a laxative. Golytely is approved by the FDA for this purpose. Another laxative, called MiraLax, is approved by the FDA to relieve constipation, but it is not approved specifically for preparation for a colonoscopy. Nonetheless, it is commonly used in clinical practice for this purpose, just as is Golytely. The purpose of this study is to compare Golytely and MiraLax in two ways: to see whether one is better tolerated by patients than the other and to see whether one more effectively cleanses the bowel than the other. The investigators' hypothesis is that these 2 bowel preparation methods are equally effective in bowel cleansing, but that patients prefer Miralax to Golytely.

ELIGIBILITY:
Inclusion Criteria:

* average risk screening for colon cancer

Exclusion Criteria:

* subjects with a history of constipation

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
bowel cleanliness as rated by the boston bowel prep survey | measured at the time of colonoscopy

SECONDARY OUTCOMES:
patient tolerability | measured at check in to colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Sciences University, Portland, Oregon, United States

REFERENCES:
- [Derived] Enestvedt BK, Fennerty MB, Eisen GM. Randomised clinical trial: MiraLAX vs. Golytely - a controlled study of efficacy and patient tolerability in bowel preparation for colonoscopy. Aliment Pharmacol Ther. 2011 Jan;33(1):33-40. doi: 10.1111/j.1365-2036.2010.04493.x. Epub 2010 Oct 25. PMID 21083586